CLINICAL TRIAL: NCT03286608
Title: Pattern of Polyphenol Intake and the Long-term Risk of Dementia in Older Persons
Brief Title: Polyphenols and Risk of Dementia
Status: Completed | Type: Observational
Sponsor: Jean-François Dartigues (Other)
Responsible Party: Sponsor-Investigator, Jean-François Dartigues, Pr, University of Bordeaux
Organization: University of Bordeaux (Other)
Other Study IDs: Three-City study Bordeaux
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Diet, Polyphenols, Flavonoids, Stilbenes, Aged, Dementia, Alzheimer's Disease, Epidemiology
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study (no intervention) — Statistical association between adherence to a pattern of polyphenol intake and the risk to develop dementia and Alzheimer's disease over 12 years
  Other Names: pattern of polyphenol intake

SUMMARY:
This project aims to leverage existing data from a large observational prospective study on dementia, the Three-City study, to investigate the relationship between intakes of polyphenols and the risk to develop dementia in the 12 years following dietary assessment.

DETAILED DESCRIPTION:
The study sample includes 1,329 subjects followed for up to 12 years fro dementia after dietary assessment. The aim is to identify a pattern of polyphenol intake (based on 26 flavonoid and non-flavonoid polyphenol subclasses ascertained using a 24-hour dietary recall) associated with the risk of dementia and AD over 12 years in the 3C Bordeaux cohort.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or more, live in Bordeaux area (France)

Exclusion Criteria:

* with dementia at the time of dietary assessment in year 2001-2002

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: population of older persons from the community, aged 65 years or more, living in the Bordeaux area (France)
Sampling Method: Non-Probability Sample
Enrollment: 1329 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of dementia | 12 years
  incident cases of dementia diagnosed by the expert committee of neurologists at follow-up visits

SECONDARY OUTCOMES:
incidence of Alzheimer's disease | 12 years
  dementia with probable or possible Alzheimer etiology

IPD SHARING:
Plan to Share IPD: No